CLINICAL TRIAL: NCT03104569
Title: Effect of 37℃ Non-ionic Contrast Agent During ERCP Procedure in Hilar Cholangiocarcinoma: A Prospective Double-blind Multicenter Randomized Controlled Study
Brief Title: Effect of 37℃ Non-ionic Contrast Agent During ERCP Procedure in Hilar Cholangiocarcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Xun Li, M.D., Ph. D, Director., Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 37℃ Contrast Agent in ERCP
Record Dates: First submitted 2017-03-26; First posted 2017-04-07 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cholangitis
Keywords: ERCP; Contrast agent; Hilar cholangiocarcinoma; Cholangitis; Nonionic
MeSH Terms: conditions — Cholangitis; Klatskin Tumor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection of 37℃ contrast agent (Experimental): Nonionic contrast agent is heated to 37℃ during ERCP when injection of contrast agent
  Interventions: Procedure: Injection of 37℃ contrast agent
- Injection of normal contrast agent (No Intervention): Normal temperature nonionic contrast agent can be used in ERCP when injection of contrast agent

INTERVENTIONS:
Procedure: Injection of 37℃ contrast agent — Nonionic contrast agent is heated to 37℃ in a incubator when injection of contrast agent
  Arms: Injection of 37℃ contrast agent

SUMMARY:
The purpose of this study is to determine the effect of normal temperature and 37℃ non-ionic contrast agent acting on ERCP-related cholangeitis after endoscopic retrograde cholangiopancreatography (ERCP) in the treatment of hilar cholangiocarcinoma.

DETAILED DESCRIPTION:
At present, the common used contrast agent in ERCP is composed of ionic and non-ionic type, and the latter's advantages lie in its slighter toxic-and-side effect and favorable security. When heated to 37℃, the 20 ℃ contrast agents would be diluted to 50% consistency, then a shorter time period of its intravascular and other intracavitary stay would add to less cell damage. And the applications of heated non-ionic contrast agents could be found in computed tomography angiography(CTA), hysterosalpingography (HSG) and cystourethrography, and consequently the patients with the intervention of heated non-ionic contrast agents felt more comfortable and fewer adverse reactions could be observed. Nevertheless, heated contrast agent was rarely reported to act in ERCP. It's theoretically possible that its heat-reduced lower mucosity could help the contrast agent itself to drainage, so that the incidence of cholangeitis could be under control.

ELIGIBILITY:
Inclusion Criteria:

* Type Ⅰ、Ⅱ、Ⅲ、Ⅳ of Hilar Cholangiocarcinoma;
* Age: 18~90 years old;
* Underwent diagnostic and therapeutic ERCP;

Exclusion Criteria:

* Coagulation dysfunction(INR>1.3) or/and low peripheral blood platelet count （PLT <50x10^9/L）;
* Preoperative acute cholangitis;
* Preoperative acute pancreatitis;
* Preoperative hemobilia or hemorrhage of digestive tract;
* Preoperative liver failure;
* Combined with Mirizzi syndrome and intrahepatic bile duct stones;
* Preoperative malignant tumor of biliary system such as carcinoma of head of pancreas, gallbladder carcinoma;
* Biliary-duodenal fistula confirmed during ERCP;
* A history of reconstructive surgery for upper digestive tract except Billroth Ⅰand a history of cholangioenterostomy including cholangio-jejunostomy and side to side anastomosis of the bile duct and duodenum;
* Previous ERCP;
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Acute cholangitis | 2 weeks
  Acute cholangitis is defined if patients experienced abdominal pain, high fever(over 38.5℃), or chill after procedure in 2 weeks

SECONDARY OUTCOMES:
The ease of injection | During procedures
  The ease of contrast agent injection has been considered by ERCP assistant, a questionnaire is required to assign by the assistant
Number of Participants With Abnormal Laboratory Values | 4 days
  9 parameter will be collected in day 2 and day 4 after procedures. Abnormal in Total bilirubin (TBIL), White Blood Count (WBC), N%,Platelet( PLT), Procalcitonin(PCT) or C-reactive protein(CRP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and Gamma - glutamyl transpeptidase (GGT) required to be documented
Operation time | intraoperative
  Total time of procedure
X-ray exposure time | intraoperative
  The total time of X-ray exposure
Number of participants with Post-ERCP pancreatitis | 1 months
  Post-ERCP pancreatitis is defined if patients experienced abdominal pain for more than 24h after ERCP, accompanying with amylase or lipase more than 3 times equal to the upper limit of normal value.

CONTACTS AND LOCATIONS:
Overall Officials: Xun Li, M.D., Ph. D., Study Chair — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (3):
- China (3):
  - The first hospital of Lanzhou university, Lanzhou, Gansu
  - The first affiliated hospital of Xi 'an jiaotong university, Xi'an, Shaanxi
  - Tianjin Nankai Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No